CLINICAL TRIAL: NCT06214026
Title: The Effectiveness of Frontal Plane Adaptability in a Novel Foot Prosthesis for People With Above-Knee Amputations, Bilateral Amputations, or Limited Mobility
Brief Title: Effectiveness of Frontal Plane Adaptability in a Novel Foot Prosthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Murray Maitland, Professor-Associate: Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017239; OP220033 (Other Grant/Funding Number: Department of the Army)
Record Dates: First submitted 2023-11-20; First posted 2024-01-19 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Amputation
Keywords: prosthesis; foot prosthesis; Above-knee amputation; Bilateral lower extremity amputation; mobility disability

STUDY DESIGN:
Intervention Model Description: A1, B1, B2, A2 crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Locked ankle articulation (Experimental): The design is a randomized cross-over clinical trial following an A1-B1-B2-A2 design. In the locked condition, the 20 degree of frontal plane ankle motion is eliminated by a physical lock. The A conditions will be with the usual foot. The B conditions are randomized to the locked and unlocked investigational foot.
  Interventions: Device: META-Arc foot locked
- Unlocked ankle articulation (Experimental): The design is a randomized cross-over clinical trial following an A1-B1-B2-A2 design. In the unlocked condition, the 20 degree of frontal plane ankle motion is enabled. The A conditions will be with the usual foot. The B conditions are randomized to the locked and unlocked investigational foot.
  Interventions: Device: META-Arc foot unlocked

INTERVENTIONS:
Device: META-Arc foot locked — Participants are provided with the META-Arc from WIllowWood Global, and a locking mechanism prevents side-to-side motion.
  Arms: Locked ankle articulation
Device: META-Arc foot unlocked — Participants are provided with the META-Arc from WIllowWood Global allowing side-to-side motion.
  Arms: Unlocked ankle articulation

SUMMARY:
People with lower extremity amputation (LEA) have persistent problems with balance, falls, residual limb pain, functional mobility, cognitive attention during gait, and satisfaction with participation in daily activities, despite using prostheses. The purpose of this randomized clinical trial is to advance understanding of how dynamic foot design features may help people with LEA This study will include people with above-knee amputations, or with bilateral amputations, or with below-knee amputations and lower levels of mobility.

The main study questions/goals are:

1a) To determine if frontal plane adaptation in a foot prosthesis impacts performance, comfort, activities of daily living, and community mobility in the study populations. To answer this question, we will compare a locked and unlocked version of the novel prosthesis.

1b) To determine how the unlocked investigational foot condition compares to the person's usual foot using the outcomes listed above.

2) To examine the participants' lived experience during community activities. The study will use performance tests, questionnaires, logbooks, and interviews to monitor person-centered outcomes and perceptions of personal functioning during the use of the investigational foot (locked and unlocked) compared to the person's usual foot.

DETAILED DESCRIPTION:
The study design is a randomized cross-over clinical trial design (B1 and B2 phases) comparing a carbon fiber foot that includes a functional, unlocked frontal plane adaptable linkage compared to the same foot with the linkage locked to prevent frontal plane motion. With the linkage locked, the foot is comparable to energy storage and return of a carbon fiber foot. The secondary aim for this clinical trial compares the unlocked foot to the participant's usual foot (A1 and A2 phases), representative of the usual standard of care.

The testing will be conducted following an A1-B1-B2-A2 design. The A conditions are focused on the participant's usual prosthetic foot. The B conditions are focused on locked and unlocked frontal plane adaptable linkages with the order randomized. Block randomization, stratified by study site, will be used to determine the order participants receive the locked and unlocked prosthetic. In our recent clinical trial, we developed a simple pin system to prevent the linkage from rotating.

A1 represents Visit 1, where demographic data are entered. As well, baseline questionnaires and performance data are collected. The participant will become familiar with the online data gathering systems. Then, the participant will be fitted with the adaptable foot by a licensed prosthetist. The linkage will be either locked or unlocked depending on the randomization. People with bilateral amputations will receive symmetrical prostheses.

During the ~2-week B1 phase, the participant will perform their normal community activities and contribute usage data, performance ratings, and qualitative data via the online logbook. There is the possibility that the decision may be made to re-fit the participant with a different stiffness of the study foot/feet that will be better suited. If this happens, the at-home use period of participation will be extended for another 2- to 4 weeks. At the end of the B1 phase, participants will complete standardized questionnaires and performance tests at Visit 2. Then, the linkage will be either locked or unlocked depending on the B1 randomization.

The ~2-week B2 phase will allow the participant to continue community activities and complete online logbooks. At the finish of the B2 phase, questionnaires and performance tests will be completed at Visit 3. A semi-structured interview will occur to compare the locked and unlocked versions.

The purpose of the second ~2-week A2 phase is for the participant to reflect on differences between the adaptable foot and the usual foot after having experiences with the adaptable linkage in the unlocked configuration. Questionnaires and an interview will occur at the final participant session, Visit 4.

Questionnaires: The demographic survey, online questionnaires, and activity logbooks will be developed in REDCap and administered either online or on paper, depending on the participant's preferences. Unique URL invitations are sent to participants via email, and reminders are sent if there is a delay in data entry. Data are collected in a database format for analysis.

Demographic questions cover age, gender, date of amputation, number of prosthetic feet, description of the usual foot (feet), walking aids, overall health rating, fall history, occupation (if working), physical activity, comorbidities, amputation etiology, veteran status, employment status, education level, race, and ethnicity.

The Prosthetic Limb Users Survey of Mobility (PLUS-M™) The PLUS-M 12-item questionnaire examines the difficulty of typical everyday mobility activities on a 5-point Likert scale.

Logbooks: Participants will complete daily structured logbooks. Daily logbooks will capture information about prosthetic use (which prosthesis was worn, length of time worn), any falls, residual limb/bodily pain, and provide an opportunity to make notes about any activities that were noticeably impacted by the prosthetic foot. There will be opportunities for participants to provide information about challenging situations and social interaction using scales and open-ended questions. Participants will be encouraged to provide descriptions of activities, including strengths and limitations of foot performance, and to address ADL that might be associated with secondary conditions such as pain, poor balance, safety, fear of falling, attention to foot placement, bilateral activities, surfaces, and uneven ground. Logbooks will be developed in REDCap and can be completed online or on paper. Logbook data will inform the content of the interviews.

Semi-structured Interviews: There will be interviews after research phases B2 (innovative foot) and A2 (usual foot). These interviews will clarify significant events documented in the logbooks. The focus of interviews will be on gathering information about the participants' experience using different prosthetic feet, with an emphasis on identifying activities that are facilitated or hindered by the functioning of the prosthetic foot. Interviews will be audio recorded for transcription and analysis.

Physical performance tests Forward walking (10-meter walk test) Forward walking at a self-selected speed is a basic test of mobility and is correlated to community function. Spatiotemporal variables during this test will be measured using an instrumented Zeno Walkway.

The Timed Up and Go Test (TUG) For the TUG, the participant, starts sitting in a chair and, on the command "go," rises, walks 3 meters, turns 180 degrees, returns to the chair, and sits down. There is typically one practice and one test. This is a timed test. In addition to total time, spatiotemporal variables during the TUG will be collected using an instrumented Zeno Walkway.

The Three Times Figure of Eight Walk Test (3XF8W) The 3XF8W involves significant turning requirements for the participant. The test was developed to represent walking skills used in everyday life, involving straight and curved paths in both right and left directions. Subjects will begin the task standing between the 2 cones 1.52 m apart. The subject will walk a figure 8 course 3 times for each condition at their self-selected pace and stop when they return to the start position. The outcomes of the test are the time to complete the course and the number of steps taken.

Four-square step test (FSST) The FSST is a complex stepping sequence. The participant is instructed to "Try to complete the sequence as fast as possible without touching the sticks. Both feet must contact the floor in each square. If possible, face forward during the entire sequence." The performance tests are ordered in increasing complexity and challenge for people with lower levels of mobility. The FSST combines side-step in both directions, as well as forward and backward stepping. Spatiotemporal variables during this test will also be collected on an instrumented Zeno Walkway.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 16-years or older, regardless of gender, race, or ethnicity.
* Potential participants should reside in the community or an independent living environment.
* The upper weight limit is 165.6 kg (365 lbs.).
* Prosthetic foot sizes 22 cm (approximate US Men's shoe size 5) up to 30 cm (13 US Men's).
* Ability to walk more than 400 m on level ground without an increase in pain.
* At least one year post-amputation and using a prosthesis
* People must have the ability to read, write, and comprehend English.

Exclusion Criteria:

* Participants must not have conditions such as skin wounds that preclude the use of a prosthesis.
* People will be excluded if they have fluctuating conditions that may significantly alter gait mechanics during the ~10-week study. Examples include Parkinson's disease, alcoholism, brain tumor, and hereditary cerebellar ataxias.
* Participants may use a walking aid but should not primarily rely on wheelchair mobility.
* People will be discontinued from the study if they become unable to use a prosthesis. Examples include major surgery and trauma. However, because of the potential for fluctuations in prosthesis use with this population, short-term issues will not disqualify people from continued participation when they resume prosthetic use.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  Forward walking for 10 meters at a self-selected speed.
Timed Up and Go Test | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  The Timed Up and Go Test starts with participant sitting in a chair. On the command "go," the individual will get up and walk 3 meters, turn 180 degrees to walk back the way they came, return to the chair, and sit down. There is one practice and one test.
Figure-of-8 Walk Test | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  For the Figure-of-8 Walk Test the participant will walk at their own pace three times in a figure-of-8 pattern around two cones placed 5 feet apart. They will have the opportunity to practice, and then the test will be repeated three times.
The Four-square Step Test (FSST) | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  The Four-square Step Test (FSST) involves stepping sideways, backwards, and forward following a pattern.
The Prosthetic Limb Users Survey of Mobility (PLUS-M™) | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  The PLUS-M 12-item questionnaire examines typical everyday mobility activities on a 5-point Likert scale.

SECONDARY OUTCOMES:
Spatiotemporal parameters of gait | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  Degree of asymmetry: Percent difference
Spatiotemporal parameters of gait | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  Step width: meters
Spatiotemporal parameters of gait | After 2-week trial of investigational foot Condition 1 (B1), after 2-week trial of investigational foot Condition 2 (B2) after return to usual foot for 2 weeks (A2).
  Step length: meters
Daily Activity Logbook: Balance Confidence | Average of daily logbook across the 2-week trial of each investigational foot condition.
  Self-reported confidence in balance on a 0-100 scale (higher scores indicate greater confidence).

CONTACTS AND LOCATIONS:
Overall Officials: Murray Maitland, PT, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of South Florida, Tampa, Florida
  - WillowWood Global, Mount Sterling, Ohio
  - University of Washington, Seattle, Washington